CLINICAL TRIAL: NCT05260138
Title: Effect of Massaging on Bilirubin Level Among Full Term Neonates With Hyperbilirubinemia Under Phototherapy.
Brief Title: Bundling Gentle Body Massage Along With Regular Position Change Under Phototherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Zohour Ibrahim Mahmoud Rashwan, Lecturer, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 170301221
Record Dates: First submitted 2022-02-18; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Hyperbilirubinemia, Neonatal
Keywords: Hyperbilirubinemia; neonatal; Massage Therapy; Bilirubin; Stool frequency; Length of Hospital Stay
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal; Hyperbilirubinemia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The intervention group (Experimental): received all basic routine care in addition to regular position change and gentle body massage
  Interventions: Other: Gentle Body message
- The control group (Active Comparator): received the conventional NICU care
  Interventions: Other: Routine NICU Care

INTERVENTIONS:
Other: Gentle Body message — The intervention group received gentle body massage twice/day and position change from supine to lateral every two hours under the phototherapy for three consecutive days in addition to routine NICU care.
  Arms: The intervention group
Other: Routine NICU Care — received the conventional NICU care of infants undergoing phototherapy. Phototherapy was given by single Blue LEDs emitting light in a narrow spectrum (450-470 nm). Initially, phototherapy lamps were checked and adjusted at the height of 30 cm from the neonates who were kept naked in the incubator/crib except for the reproductive organs with shielded eyes. The neonates were positioned supine under the phototherapy. The treatment was given continuously, except while feeding and nursing for 30 minutes every 3 hours. The neonates' skin was cleaned with warm water without applying any sorts of ointments oils or creams. They were also observed for signs of dehydration.
  Arms: The control group

SUMMARY:
This study aimed to investigate the effect of bundling gentle body massage along with regular position change on bilirubin level and clinical outcomes among full-term neonates with hyperbilirubinemia under phototherapy.

Hypothesis

Full-term neonates with hyperbilirubinemia who receive gentle body massage along with regular position change exhibit less bilirubin level and better clinical outcomes than those who don't.

DETAILED DESCRIPTION:
A quasi-experimental study was carried out in the NICU of XX. Sixty full-term neonates were randomly assigned to two equal groups.

The control group received the conventional NICU care of infants undergoing phototherapy. Phototherapy was given by single Blue LEDs emitting light in a narrow spectrum (450-470 nm). Initially, phototherapy lamps were checked and adjusted at the height of 30 cm from the neonates who were kept naked in the incubator/crib except for the reproductive organs with shielded eyes. The neonates were positioned supine under the phototherapy. The treatment was given continuously, except while feeding and nursing for 30 minutes every 3 hours. The neonates' skin was cleaned with warm water without applying any sorts of ointments oils or creams. They were also observed for signs of dehydration.

The intervention group received all basic routine care in addition to regular position change from supine to laterals under the phototherapy every two hours. They also received gentle body massage

ELIGIBILITY:
Inclusion Criteria:

* Full-term
* receive enteral feeding (breast, bottle, or mixed feeding, gavage)
* Newly admitted

Exclusion Criteria:

* Required exchange transfusion
* Required mechanical ventilation
* Has acute phase of circulatory insufficiency
* Hemolytic disease
* Neurological disorders
* Congenital anomalies
* Neonatal sepsis Diarrhea

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2021-08-20 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2021-12-18 (Actual)

PRIMARY OUTCOMES:
Bilirubin level | After 3 days
  The researchers recorded the neonates' Bilirubin level from the laboratory results

SECONDARY OUTCOMES:
Percentage of the consumed milk | After 3 days
  The researchers calculated the percentage of the consumed milk by dividing the actual amount sucked by the neonate on the prescribed amount and multiplied by 100
Frequency of stool | After 3 days
  The researchers counted number of neonates' stool passage per day
daily weight | After 3 days
  The researchers measured the neonates' weight daily using the same scale
Length of hospital stay | After 10 days
  the researchers obtained the neonates' length of hospital stay from admission to discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang M, Wang L, Wang Y, Tang J. The influence of massage on neonatal hyperbilirubinemia: a meta-analysis of randomized controlled trials. J Matern Fetal Neonatal Med. 2019 Sep;32(18):3109-3114. doi: 10.1080/14767058.2018.1455183. Epub 2018 Apr 9. PMID 29631455
- [Background] Chen A, Du L, Xu Y, Chen L, Wu Y. The effect of blue light exposure on the expression of circadian genes: bmal1 and cryptochrome 1 in peripheral blood mononuclear cells of jaundiced neonates. Pediatr Res. 2005 Dec;58(6):1180-4. doi: 10.1203/01.pdr.0000183663.98446.05. PMID 16306190
- [Background] Donneborg ML, Knudsen KB, Ebbesen F. Effect of infants' position on serum bilirubin level during conventional phototherapy. Acta Paediatr. 2010 Aug;99(8):1131-4. doi: 10.1111/j.1651-2227.2010.01885.x. Epub 2010 Jun 2. PMID 20528799
- [Background] Field TM, Schanberg SM, Scafidi F, Bauer CR, Vega-Lahr N, Garcia R, Nystrom J, Kuhn CM. Tactile/kinesthetic stimulation effects on preterm neonates. Pediatrics. 1986 May;77(5):654-8. PMID 3754633
- [Background] Kato S, Iwata O, Yamada Y, Kakita H, Yamada T, Nakashima H, Sugiura T, Suzuki S, Togari H. Standardization of phototherapy for neonatal hyperbilirubinemia using multiple-wavelength irradiance integration. Pediatr Neonatol. 2020 Feb;61(1):100-105. doi: 10.1016/j.pedneo.2019.07.002. Epub 2019 Aug 12. PMID 31473126